CLINICAL TRIAL: NCT00126971
Title: Pharmacokinetics of Chlorproguanil-Dapsone in Pregnant Women With Plasmodium Falciparum Infection, and Reinfection With P. Falciparum During Pregnancy Following Treatment
Brief Title: Chlorproguanil-Dapsone in Pregnant Women
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); Liverpool School of Tropical Medicine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCID-4341
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Malaria
Keywords: malaria; pregnancy; Plasmodium falciparum; antimalarials; pharmacokinetics; treatment outcome; safety
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — chloroguanil, dapsone drug combination

INTERVENTIONS:
Drug: chlorproguanil-dapsone

SUMMARY:
Controlling malaria during pregnancy is a vital strategy in decreasing maternal and child mortality in Africa. There are data from clinical trials and program evaluations in stable transmission areas that show that intermittent preventive treatment (IPT) with two doses of sulfadoxine-pyrimethamine (SP) is safe, efficacious, and effective in preventing maternal anemia, placental parasitemia, and low birth weight (LBW). SP is also the first-line drug for the case-management of malaria in pregnancy. Resistance to SP, however, is increasing rapidly in East and Central Africa and compliance to the rescue treatment, 7-days of oral quinine, is low. There is an urgent need to find effective, safe and practical alternative drugs for the treatment of malaria in pregnancy. The synergistic antifolate combination chlorproguanil-dapsone (CD), has recently become available. It is inexpensive, well tolerated, is given as single daily treatment doses for 3 days, and is effective in the treatment of drug-resistant falciparum malaria.

The investigators propose a small pharmacokinetic study of CD to determine if current fixed combination CD tablets provide an adequate dosage in pregnancy. Such a study is a necessary precursor to any large Phase II trials to further evaluate the safety and efficacy of CD for use in pregnant women. To accomplish this, a group of 66 parasitemic pregnant women in this open label trial will receive CD and be sampled by venipuncture at two of the seven follow-up visits scheduled for pharmacokinetic analyses, such that 11 patients are sampled at each of 12 time points. To serve as a reference, 66 non-pregnant women with symptomatic malaria will also be treated with CD and will have identical pharmacokinetic (PK) analyses performed.

Pregnant women greater than or equal to 20 weeks gestation with P. falciparum parasitemia on peripheral blood film will be given an insecticide-treated net (ITN) and will receive CD (1.5 or 2 tablets daily for 3 days, depending on weight). All study drug dosing will be observed. Women will be examined, adverse events recorded, and blood samples collected at days 0, 1, 2, 3, 7, 14, 21, and 28 after treatment, and thereafter every 14 days until delivery. Women will be further randomized to receive additional blood draws for pharmacokinetic analyses using a modified rich PK schedule. Each woman will only have 2 additional blood draws. Women at delivery will have peripheral and placental blood films prepared. Newborns will be weighed, examined, and gestational age determined. Women requiring antimalarial treatment for parasitemia at any point between enrollment and delivery will be treated with quinine. Adverse effects will be assessed at each scheduled visit, any sick visits during the study, and at delivery.

DETAILED DESCRIPTION:
Malaria infection during pregnancy poses substantial risk to the mother, her fetus, and the neonate. In areas of stable transmission where adult women have considerable acquired immunity, Plasmodium falciparum infection during pregnancy typically does not cause symptomatic malaria, but may lead to maternal anemia and placental malaria infection, especially among primigravidae and secundigravidae. This placental malarial infection contributes to low birth weight (LBW), a major contributor to infant mortality. Malaria contributes up to 15% of maternal anemia, 14% of LBW, 30% of preventable LBW, 70% of intrauterine growth retardation, 36% of premature delivery, and 8% of infant mortality. In Mali, malaria is the leading cause of morbidity (15%) and mortality (13%) in the general population (Kassoum Kayentao, personal communication). Malaria can be found in 25.9% of pregnant women attending antenatal care, and in the placenta of 27.8% of pregnant women at delivery (Kassoum Kayentao, personal communication).

Controlling malaria during pregnancy is a vital strategy in decreasing maternal and child mortality in Africa. There are data from clinical trials and program evaluations in stable transmission areas that show that intermittent preventive treatment (IPT) with two doses of sulfadoxine-pyrimethamine (SP) is safe, efficacious, and effective in preventing maternal anemia, placental parasitemia, and LBW. SP is also the first-line drug for the case-management of malaria in pregnancy. Resistance to SP, however, is increasing rapidly in East and Central Africa and compliance to the rescue treatment, 7-days of oral quinine, is low. There is an urgent need to find effective, safe and practical alternative drugs for the treatment of malaria in pregnancy. The synergistic antifolate combination chlorproguanil-dapsone (CD), has recently become available as a fixed combination caplet of 80 mg chlorproguanil and 100 mg dapsone (Lapdap™, GlaxoSmithKline, UK). It is inexpensive ($0.29 per treatment course), well tolerated, is given as single daily treatment doses for 3 days, and is effective in the treatment of drug-resistant falciparum malaria. CD however has good efficacy as salvage therapy of SP treatment failures in children and could play an important role in the case management of malaria in pregnancy. Given that the component drugs are both considered safe in pregnancy, it is expected that the combination will also be safe for use in pregnancy, but this has not been formally evaluated.

The investigators propose a small pharmacokinetic study of CD to determine if the current co-formulated fixed combination CD tablets provide an adequate dosage in pregnancy. Such a study is a necessary precursor to any large Phase II trials to further evaluate the safety and efficacy of CD for use in pregnant women. Therefore, the primary objective of this study is to evaluate the pharmacokinetics of CD in pregnancy. To accomplish this, a group of 66 parasitemic pregnant women in this open label trial will receive CD and be sampled by venipuncture at two of the seven follow-up visits scheduled for pharmacokinetic analyses, such that 11 patients are sampled at each of 12 time points. To serve as a reference, 66 non-pregnant women with symptomatic malaria will also be treated with CD and will have identical PK analyses performed.

There are also data that show that women using insecticide treated bednets (ITNs) during pregnancy are also less likely to suffer the adverse outcomes of malaria during pregnancy. The World Health Organization (WHO) currently recommends that all pregnant women in malaria endemic areas sleep under an ITN and receive at least 2 doses of IPT with an efficacious antimalarial in the 2nd and 3rd trimester. The combined efficacy of ITNs and IPT remains unclear. It is important to understand if a short-acting antimalarial such as CD will function as well as a long-acting drug such as SP in preventing malaria during pregnancy among women who are also sleeping under an ITN. Therefore, the secondary aim is to estimate the proportion of pregnant women sleeping under ITNs who become re-infected with malaria before delivery following administration of a single dose of chlorproguanil-dapsone for P. falciparum parasitemia.

Eligible pregnant women greater than or equal to 20 weeks gestation with P. falciparum parasitemia on peripheral blood film, with no history of antimalarial use other than chloroquine or quinine, and who give consent to participate will be given an ITN and will receive CD (1.5 or 2 tablets daily for 3 days, depending on weight) All study drug dosing will be observed. Women will be examined, adverse events recorded, and blood samples collected at days 0, 1, 2, 3, 7, 14, 21, and 28 after treatment, and thereafter every 14 days until delivery. Women will be further randomized to receive additional blood draws for pharmacokinetic analyses using a modified rich PK schedule. Each woman will only have 2 additional blood draws. Women at delivery will have peripheral and placental blood films prepared. Newborns will be weighed, examined, and gestational age determined. Women requiring antimalarial treatment for parasitemia at any point between enrollment and delivery will be treated with quinine. Adverse effects will be assessed at each scheduled visit, any sick visits during the study, and at delivery. An independent external monitor will be recruited for visiting the study site at the beginning of the field work and before the end of the study.

Standard pharmacokinetic measurements using high-pressure liquid chromatography will be performed to determine serum CD levels. Determination of malaria parasitemia (peripheral and placental) will be made by reading thick Giemsa-stained blood films. Birth weights will be measured using an electronic scale (+/- 10g). Gestational age will be estimated using the Ballard score. All women will receive an ITN on enrollment to reduce the probability of new malaria infections of mother and newborn.

ELIGIBILITY:
Inclusion Criteria:

For the pregnancy part of the study, a subject will be considered eligible for inclusion in this study only if all of the following criteria apply: She

* Is pregnant and presents at the antenatal clinic (ANC) facilities of the study hospital.
* Has uncomplicated malaria (either symptomatic or not) with pure (on microscopic grounds) P falciparum parasitemia.
* Has a gestational age of >= 20 and < 36 weeks (defined by fundal height).
* Is willing and able to participate and comply with the study protocol, attend the ANCs regularly and agrees to supervised drug delivery.
* Has no history of antimalarial intake in the previous 4 weeks, with the exception of chloroquine or quinine.
* Has given written or witnessed verbal consent.

For the 66 non-pregnant women, the following inclusion criteria will apply:

* Has uncomplicated malaria (either symptomatic or not) with pure (on microscopic grounds) P falciparum parasitemia.
* Negative urine pregnancy test.
* Is willing and able to participate and comply with the study protocol, attend the ANCs regularly and agrees to supervised drug delivery.
* Has no history of antimalarial intake in the previous 4 weeks, with the exception of chloroquine or quinine.
* Has given written or witnessed verbal consent.

Exclusion Criteria:

* Any feature of severe malaria.
* A history of convulsions during the present illness.
* Known history of G6PD deficiency or sickle cell disease.
* Other conditions requiring hospitalization or evidence of severe concomitant infection at time of presentation.
* Women on daily cotrimoxazole prophylaxis
* Use of any antimalarial (other than chloroquine or quinine) in the past 4 weeks.
* Known chronic disease (cardiac, renal, hepatic, hemoglobinopathy), or known hepatic or renal impairment.
* Inability to follow the ANC consultation.
* Hemoglobin < 7 g/dL (will be measured before enrollment)
* Inability to tolerate oral treatment reflected by persistent vomiting of the study drugs.
* Known allergy to either the study drugs, or to any sulfa-containing medications.
* Age <15 years.
* Age >49 years.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2005-07

PRIMARY OUTCOMES:
Pharmacokinetic analyses of pregnant women taking CD

SECONDARY OUTCOMES:
Proportion of pregnant women sleeping under ITNs who become re-infected with malaria before delivery following administration of a single dose of CD for P. falciparum parasitemia
Proportion of treatment failures by day 28 following initial treatment
Treatment failure will be defined according to standard WHO criteria for low to moderate transmission areas to account for fact that some pregnant women are asymptomatic
Early treatment failure: development of danger signs or severe malaria on Day 1, Day 2 or Day 3 in the presence of parasitemia (severe malaria defined by altered sensorium convulsions
persistent vomiting
renal impairment
respiratory distress)
a fall in Hb below 5g/dl anytime
parasitemia on Day 2 higher than Day 0 count irrespective of axillary temperature
parasitemia on Day 3 with axillary temperature >= 37.5 °C
parasitemia on Day 3 >= 25% of count on Day 0
Late clinical failure: development of danger signs of severe malaria after Day 3 in the presence of parasitemia, without previously meeting any of the criteria of early treatment failure
presence of parasitemia and axillary temperature >= 37.5 °C on any day from Day 4 (inclusive) to Day 28 (inclusive), without previously meeting any of the criteria of early treatment failure
Late parasitological failure: parasitemia on any day between Day 7 (inclusive) and Day 28 (inclusive)
axillary temperature <37.5 °C without previously meeting any of the criteria of early treatment failure or late clinical failure, after exclusion of re-infection by PCR (days
adequate clinical and parasitological response [ACPR] will be defined as: absence of parasitemia on Day 28 irrespective of axillary temperature without previously meeting any of the criteria of early treatment failure
or late clinical failure
or late parasitologic failure)
Parasite clearance by Day 3
Mean Hb concentrations by Day 28, and hematological recovery by day 28 (Hb > 11 g/dL)
Gametocytemia
Maternal parasitemia at delivery
Placental malaria parasitemia
Mean birth weight and gestational age of newborn
Presence of congenital abnormalities
Incidence of fetal loss
Incidence of perinatal and neonatal mortality, assessed 4-6 weeks after due date of delivery
Incidence of fetal death, defined as absence of fetal heartbeat
Hypoglycemia requiring treatment
Other adverse events during treatment period (up to 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Newman, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Kassoum Kayentao, MD, MSPH, Principal Investigator — Malaria Research and Training Center; Feiko ter Kuile, MD, PhD, Principal Investigator — Liverpool School of Tropical Medicine; Ogobara Doumbo, MD, PhD, Principal Investigator — Malaria Research and Training Center; Monica E Parise, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Faladje Missionary Dispensary, Faladié, Mali

REFERENCES:
- [Background] Mutabingwa T, Nzila A, Mberu E, Nduati E, Winstanley P, Hills E, Watkins W. Chlorproguanil-dapsone for treatment of drug-resistant falciparum malaria in Tanzania. Lancet. 2001 Oct 13;358(9289):1218-23. doi: 10.1016/S0140-6736(01)06344-9. PMID 11675058
- [Background] Keuter M, van Eijk A, Hoogstrate M, Raasveld M, van de Ree M, Ngwawe WA, Watkins WM, Were JB, Brandling-Bennett AD. Comparison of chloroquine, pyrimethamine and sulfadoxine, and chlorproguanil and dapsone as treatment for falciparum malaria in pregnant and non-pregnant women, Kakamega District, Kenya. BMJ. 1990 Sep 8;301(6750):466-70. doi: 10.1136/bmj.301.6750.466. PMID 2207399
- [Background] Winstanley P, Watkins W, Muhia D, Szwandt S, Amukoye E, Marsh K. Chlorproguanil/dapsone for uncomplicated Plasmodium falciparum malaria in young children: pharmacokinetics and therapeutic range. Trans R Soc Trop Med Hyg. 1997 May-Jun;91(3):322-7. doi: 10.1016/s0035-9203(97)90093-6. PMID 9231209